CLINICAL TRIAL: NCT02065739
Title: A Study to Investigate the Potential Effects of Repeated Administration of Itraconazole on the Pharmacokinetics of JNJ-42165279 in Healthy Male Subjects
Brief Title: A Study to Investigate the Effects of Itraconazole on the Pharmacokinetics of JNJ-42165279 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103432; 42165279EDI1004 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Healthy; JNJ-42165279; Itraconazole; Pharmacokinetics
MeSH Terms: interventions — JNJ-42165279; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): Participants will receive a single 30-mg dose of JNJ-42165279 on Day 1.
  Interventions: Drug: JNJ-42165279
- Period 2 (Experimental): Participants will receive itraconazole 200 mg once a day from Day 4 to Day 10. A single oral 30-mg dose of JNJ-42165279 will be administered on Day 8 along with the dose of 200 mg itraconazole.
  Interventions: Drug: JNJ-42165279; Drug: Itraconazole

INTERVENTIONS:
Drug: JNJ-42165279 — Participants will receive a single 30-mg (6 mL of oral suspension) dose of JNJ-42165279 orally (by mouth) on Day 1 (Period 1) and on Day 8 (Period 2).
Drug: Itraconazole — Participants will receive itraconazole 200 mg (2 capsules) once a day orally on Days 4, 5, 6, 7, 8, 9, and 10 (Period 2).
  Arms: Period 2

SUMMARY:
The purpose of this study is to assess the effects of repeated administration of 200 mg of itraconazole on the single-dose pharmacokinetics of JNJ-42165279 in healthy male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), study in healthy male participants. This study will consist of a screening phase (between 21 and 2 days prior to the first dose administration of JNJ-42165279), a 2-period (Period 1: Day 1 to Day 3 and Period 2: Day 4 to Day 10) open-label treatment phase, and a follow-up phase (within 7 to 14 days after the last dose of JNJ-42165279). A single 30-mg dose of JNJ-42165279 will be administered on Day 1 of Period 1. During Period 2, the administration of oral itraconazole 200 mg once a day will start on Day 4. A second single oral 30-mg dose of JNJ-42165279 will be administered on Day 8 together with the dose of 200 mg itraconazole. Sixteen healthy participants will be enrolled in this study. Safety assessments will include assessment of adverse events, supine vital signs, 12-lead electrocardiogram, clinical laboratory testing and physical examinations. The maximum study duration for each participant will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2 inclusive (BMI = weight/height2)
* Nonsmoker (not smoked for 3 months prior to screening)
* During the study and for 3 months after receiving study medication, must agree to use an adequate contraception method (eg, vasectomy, double-barrier, partner using effective contraception), always use a condom during sexual intercourse and to not donate sperm
* Participants must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission
* Clinically significant abnormal physical examination, vital signs or 12-lead electrocardiogram at screening or on Day 1, predose
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection. History of epilepsy or fits or unexplained black-outs
* Drinks, on average, more than 8 cups (more than or equal to 150 mL) of caffeine containing beverages per day
* Clinically significant acute illness within 7 days prior to study drug administration
* Has a contraindication to the use of itraconazole or any antifungal azoles

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  The Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUCt) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  AUCt is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity])of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Terminal Rate Constant (Lambda[z]) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  Lambda(z) is defined as terminal rate-constant which reflect the speed of drug elimination in vivo (within the living), and is estimated by log-linear regression analysis of the terminal phase of the plasma concentration versus time curve for at least 3 points.
Elimination Half-Life Period (T1/2) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  The Elimination Half-Life Period (T1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Relative Bioavailability (Frel) of JNJ-42165279 | Day 1 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 2 (24, 36 hours), Day 3, Day 4, Day 8 (Pre-dose and post-dose 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 16, hours), Day 9 (24, 36 hours), Day 10, and Day 11
  Relative bioavailability is the percentage of the administered dose that is systemically available.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Week 7

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- Merksem, Belgium